CLINICAL TRIAL: NCT06878755
Title: A Randomized Controlled Trial to Evaluate a Digital Sexual Assertiveness Intervention for Adolescent Sexual Minority Males
Brief Title: Evaluating a Digital Sexual Assertiveness Intervention for ASMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Eric R. Walsh-Buhi, Professor Applied Health Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20740
Record Dates: First submitted 2024-12-23; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Condomless Sex; Sexual Assault
Keywords: online intervention; digital health; sexual consent; condom use; condom negotiation; LGBTQ health; adolescents
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Intervention Model Description: PACT (Promoting Assertive Communication among Teens) is a brief online (web-based) educational program that can be taken on participants' personal devices.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Promoting Assertive Communication among Teens (PACT) (Experimental): A 30-minute digital program designed to teach adolescent sexual minority males information and skills regarding two dimensions of sexual assertiveness: consent and condom negotiation.
  Interventions: Other: Promoting Assertive Communication among Teens (PACT)
- Healthy Minds (Active Comparator): An attention-matched digital program focused on growth mindsets and mental health, designed for a general population of adolescents.
  Interventions: Other: Healthy Minds

INTERVENTIONS:
Other: Promoting Assertive Communication among Teens (PACT) — See Arm Description
  Arms: Promoting Assertive Communication among Teens (PACT)
Other: Healthy Minds — See Arm Description
  Arms: Healthy Minds

SUMMARY:
The purpose of this study is to test the effectiveness, likability, and implementation potential of PACT, an adapted digital program to teach non-heterosexual adolescent boys about sexual consent and condom negotiation in a randomized controlled trial over 9 months.

DETAILED DESCRIPTION:
Because the PACT (Promoting Affirmative Consent among Teens) digital health intervention showed evidence of effectiveness at improving sexual consent cognitions in its first trial, and was found generally likable among adolescents, the research team has adapted the program to serve as sexual assertiveness (consent and condom negotiation) training. This adapted version is tailored to the specific needs of adolescent sexual minority males (ASMM), a population that has been historically underserved by traditional sex education while also experiencing disproportionately high rates of both sexual violence victimization and condom non-use. The evaluation of the adapted PACT program (now titled Promoting Assertive Communication among Teens) will take place in an RCT with a Type 1 effectiveness-implementation hybrid design. Surveys will be administered at pre-intervention, post-intervention, 3-month follow-up, and 9-month follow-up. The investigators will assess acceptability, implementation factors, and main and secondary outcomes related to consent and condom negotiation/use.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years old
* lives in the U.S.
* identifies as a queer teen guy or sexual minority male

Exclusion Criteria:

* younger than 14
* older than 17
* does not live in U.S.
* does not identify as a queer teen guy or sexual minority male

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants will be eligible if they consider themselves "queer teen guys." Although a large percentage of the sample will be male-assigned at birth, the investigators anticipate that the total sample will also include gender-diverse adolescents, including those who are trans boys, transmasculine, non-binary, agender, genderqueer, and gender nonconforming.
Enrollment: 300 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Condom negotiation intentions | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' likelihood of using a condom during sexual intercourse with a partner
Affirmative consent intentions | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' likelihood of 1) ensuring consent is obtained from a partner prior to sexual intercourse and 2) communicating their consent affirmatively to a partner prior to intercourse
Condom negotiation self-efficacy | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' confidence in their ability to assert their desire to use a condom with a partner (5-point likert, strongly disagree to strongly agree, higher scores = higher self-efficacy)
Affirmative consent self-efficacy | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' confidence in their ability to communicate sexual consent with a partner (4-point likert, "not at all confident" to "very confident", higher scores = higher self-efficacy)

SECONDARY OUTCOMES:
Condom use | Baseline, 3 months, 9 months
  Behavioral outcome measuring whether a condom was used for sexual intercourse
Condom negotiation | Baseline, 3 months, 9 months
  Behavioral outcome measuring discussion about condom use prior to sexual intercourse
Affirmative consent communication | Baseline, 3 months, 9 months
  Behavioral outcome measuring affirmative consent communication before and during sexual intercourse
Condom attitudes | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' beliefs about the importance of condom use (items from the Condom Attitudes scale, strongly disagree to strongly agree, higher scores = more positive attitudes)
Affirmative consent attitudes | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' beliefs about the importance of affirmative consent (items from the Sexual Consent Scale-Revised, strongly disagree to strongly agree, higher scores = more positive attitudes)
Condom norms | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' personal and perceived norms about condom use (condom norms items from the Psychosocial Scales, higher score = more positive norms)
Affirmative consent norms | Baseline, immediately post-intervention, 3 months, 9 months
  Participants' personal and perceived norms about affirmative consent (Norms items from Sexual Consent Scale-Revised, strongly disagree to strongly agree, higher scores = more positive norms)
Acceptability | Immediately post-intervention
  Participants' perceptions of the likability and usefulness of the program (items adapted from Acceptability of Intervention measure, "not at all" to "a lot", higher scores = higher acceptability)

OTHER OUTCOMES:
Dose | Immediately post-intervention
  How much of the intervention did participants complete?
Cost | Baseline
  How much does it cost to implement the intervention?

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

REFERENCES:
- [Background] Javidi H, Widman L, Maheux AJ, McCrimmon J, Evans-Paulson R, Becker W. PACT: Developing and Evaluating a Digital Sexual Consent Program for Youth. J Sex Res. 2024 Mar-Apr;61(3):466-480. doi: 10.1080/00224499.2023.2208560. Epub 2023 May 15. PMID 37186689